CLINICAL TRIAL: NCT00238043
Title: Cohort Study to Determine the Long-Term Safety and Efficacy of Biogeneric Epoetin Treatment for Renal Anemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ministry of Health, Malaysia (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT 05-17
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2005-10

CONDITIONS: Chronic Kidney Disease; End-Stage Renal Failure; Anaemia
Keywords: Biogeneric Epoetin treatment; Renal anaemia; Chronic Kidney Disease; Pure Red Blood Cell Aplasia; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Biogeneric Epoetin

SUMMARY:
The purpose of this study is to establish the long-term safety and efficacy of Biogeneric Epoetin, the attainability of therapeutic target for anaemia management, and the impact of Epoetin treatment on long-term health outcome and its cost effectiveness.

DETAILED DESCRIPTION:
This study protocol is an elaboration of the original study protocol titled "A Randomized, Multi-center, Open label trial to establish the therapeutic equivalence between Biogeneric Epoetin and Eprex and to determine the long term safety profile of Biogeneric Epoetin in patients on Hemodialysis".

In the first stage, a biogeneric Epoetin shall be evaluated by a randomized trial designed to demonstrate therapeutic equivalence (TE) versus an innovator product (Eprex), the efficacy clinical end-point being Hb at 6 to 12 weeks on treatment.

When preliminary evidence of efficacy is established from above stage 1 TE trial, the product may proceed to be evaluated in a stage 2 single group cohort study designed to establish the long term safety, with particular emphasis on surveillance for occurrence of Pure Red Cell Aplasia (PRCA) and other immunogenicity related adverse event. To establish the long term efficacy, its emphasis on the potential impact of batch to batch variation in product content and potency (bioactivity) on Hb response.

This practical trial also designed to investigate the cost-effectiveness by estimating the optimal dosage for combination of Epoetin and Iron sucrose to achieve Hb target under unconstrained prescriptionas, and hence the budgetary requirement can be estimated to meet therapeutic target in this dialysis population under various pricing scenario in the presence of generic competition.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has Chronic Kidney Disease with anaemia for which Epoetin treatment is indicated.
* Patient without known hypersensitivity to the mammalian cell-derived product or human albumin products.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2005-08; Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
To investigate the Hb levels at each every 3 months follow up visit and the incidence of lack anticipated Hb response or loss of response to Biogeneric Epoetin. To monitor the occurrence of PRCA and other immunogenicity related adverse event.

SECONDARY OUTCOMES:
Mortality, quality of life and cost during the 6 years study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dato' Dr. Zaki Morad Mohamad Zaher, MRCP, FRCP, Principal Investigator — Department of Nephrology, Kuala Lumpur Hospital
Locations (14):
- Malaysia (14):
  - Aiman Dialysis Centre, Kuala Lumpur, Kuala Lumpur
  - Ampang Putri Specialist Hospital, Kuala Lumpur, Kuala Lumpur
  - Cheras Dialysis Centre, Kuala Lumpur, Kuala Lumpur
  - Gleneagles Intan Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Pantai Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Smartcare Dialysis Centre, Kuala Lumpur, Kuala Lumpur
  - The Kidney Dialysis Centre, Kuala Lumpur, Kuala Lumpur
  - Pahang Buddhist Association, Kuantan, Pahang
  - Pusat Hemodialisis Islam Makmur, Kuantan, Pahang
  - SP Menon Dialysis Centre, Klang, Selangor
  - SP Menon Dialysis Centre, Petaling Jaya, Selangor
  - Tan Medical Renal Clinic, Petaling Jaya, Selangor
  - Klinik Pakar Dialysis, Subang Jaya, Selangor
  - Sunway Medical Centre, Subang Jaya, Selangor

REFERENCES:
- See also: the link is an academic research organisation for the trial — http://www.crc.gov.my